CLINICAL TRIAL: NCT04595929
Title: Single-center Randomized Study Evaluating of Oncological Benifits of Pressured Intraperitoneal Aerosol Chemotherapy (PIPAC) in Patients With Locally Advanced Gastric Cancer in Patients With Cyt-.
Brief Title: Oncological Benefits of Pressured Intraperitoneal Aerosol Chemotherapy (PIPAC) in Patients With T3-4 Gastric Cancer Cyt-
Acronym: GASPACCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-AbOn-2020
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-10

CONDITIONS: Peritoneal Carcinomatosis; Gastric Cancer
Keywords: Gastric cancer; Aerosol Chemotherapy; Regional Chemotherapy; Peritoneal Carcinomatosis; Peritoneal washings; Intraperitoneal chemotherapy
MeSH Terms: conditions — Peritoneal Neoplasms; Stomach Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel; Chemotherapy, Adjuvant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIPAC group (Experimental): 1. Staging laparoscopy + peritoneal lavage.
  2. 4 cycles of neoadjuvant chemotherapy: FLOT = Docetaxel 50 mg/m², Oxaliplatin 85 mg/m², Leucovorin 200 mg/m², 5-FU 2600 mg/m² every 2 weeks.
  3. Radical gastrectomy with D2 - lymph node dissection.
  4. Intraoperative Pressured Intraperitoneal Aerosol Chemotherapy (PIPAC) with cisplatin 7,5 mg/m², doxorubicin 1,5 mg/m².
  5. Adjuvant chemotherapy according to indications.
  Interventions: Procedure: Staging laparoscopy; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Docetaxel; Procedure: Radical surgery; Procedure: PIPAC; Drug: Adjuvant chemotherapy
- Control group (Active Comparator): 1. Staging laparoscopy + peritoneal lavage.
  2. 4 cycles of neoadjuvant chemotherapy: FLOT = Docetaxel 50 mg/m², Oxaliplatin 85 mg/m², Leucovorin 200 mg/m², 5-FU 2600 mg/m² every 2 weeks.
  3. Radical gastrectomy with D2 - lymph node dissection.
  4. Adjuvant chemotherapy according to indications.
  Interventions: Procedure: Staging laparoscopy; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Docetaxel; Procedure: Radical surgery; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Procedure: Staging laparoscopy — All patients undergo staging laparoscopy and peritoneal lavage.
Drug: 5-Fluorouracil — Day 1 q2w: 2600 mg/m² IV over 24 hours
  Other Names: 5-FU
Drug: Leucovorin — Day 1 q2w: 200 mg/m² IV over 30 minutes
  Other Names: Calciumfolinat
Drug: Oxaliplatin — Day 1 q2w: 85 mg/m² IV over 2 hours
Drug: Docetaxel — Day 1 q2w: 50 mg/m² IV over 1 hour
Procedure: Radical surgery — Radical gastrectomy with D2 - lymph node dissection.
Procedure: PIPAC — Intraoperative Pressured Intraperitoneal Aerosol Chemotherapy (PIPAC) with cisplatin 7,5 mg/m², doxorubicin 1,5 mg/m².
  Arms: PIPAC group
Drug: Adjuvant chemotherapy — Adjuvant chemotherapy according to indications.

SUMMARY:
Stomach cancer is recognized as the third leading cause of death of cancer patients worldwide. Despite the radical treatment carried out, the progression of gastric cancer occurs in 30-40% of patients. The most common type of tumor progression of this localization is peritoneal carcinomatosis. When peritoneal carcinomatosis occurs, the median survival of patients does not exceed 3 months, the overall survival is no more than 6 months. Unfortunately, when peritoneal carcinomatosis occurs, palliative chemotherapy remains the only treatment option. The modern strategy for the prevention and treatment of peritoneal carcinomatosis is based on the concept of regional chemotherapy. The main methods of regional chemotherapy are hyperthermic intraperitoneal chemotherapy (HIPEC) and Pressured Intraperitoneal Aerosol Chemotherapy (PIPAC). PIPAC is a new technology for delivering chemotherapy drugs to tumor nodes on the surface of the peritoneum and allows the cytostatic to be evenly distributed over the abdominal cavity, increasing the depth of its penetration into tumor nodes due to the properties of aerosol and gradients of intra-abdominal and interstitial pressure. The method has a number of advantages over the HIPEC method: a large penetration depth of drugs, low trauma, the possibility of repeated use. We offer PIPAC for patients with locally advanced gastric cancer and a high risk of developing peritoneal carcinomatosis in an adjuvant mode in addition to standard treatment to prevent the development of carcinomatosis.

DETAILED DESCRIPTION:
The study is interventional: patients over 18 years of age with an established diagnosis of stomach cancer (c)T3-4N0-3M0 CYT- will be randomized into 2 groups using the envelope method. The control group will receive only neoadjuvant chemotherapy + gastrectomy/ distal subtotal resection with D2 lymph node dissection, the active comparison group - neoadjuvant chemotherapy + gastrectomy with D2 lymph node dissection + PIPAC (Cisplatin (7.5 mg / m²) + Doxirubicin 1.5 mg / m2)). Will be assessed: overall survival, median survival, disease-free survival, quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, medically operable, resectable stomach adenocarcinoma (cT3-4, any N category, M0).
* No preceding cytotoxic or targeted therapy.
* No prior partial or complete tumor resection.
* Female and male patient ≥ 18 and ≤ 75 years. Female patient with childbearing potential needs to have a negative pregnancy test within 7 days prior to study start. Males and females of reproductive potential must agree to practice highly effective contraceptive measures* during the study. Male patients must also agree to refrain from father a child during treatment and additionally to use a condom during treatment period. Their female partner of childbearing potential must also agree to use an adequate contraceptive measure.

  *highly effective (i.e. failure rate of <1% per year when used consistently and correctly) methods: intravaginal and transdermal combined (estrogen and progestogen containing) hormonal contraception; injectable and implantable progestogen-only hormonal contraception; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence (complete abstinence is defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments).
* ECOG = 0-2.
* Exclusion of distant metastases by CT or MRI of abdomen, pelvis, and thorax, bone scan or MRI (if bone metastases are suspected due to clinical signs). Exclusion of the infiltration of any adjacent organs or structures by CT or MRI.
* Laparoscopic exclusion of peritoneal carcinomatosis at initial staging, before start of FLOT chemotherapy
* Adequate hematological, hepatic and renal function parameters:

Leukocytes ≥ 3000/mm³, platelets ≥ 100,000/mm³, neutrophil count (ANC) ≥1000/µL Serum creatinine ≤ 1.5 x upper limit of normal Bilirubin ≤ 1.5 x upper limit of normal, AST and ALT ≤ 3.0 x upper limit of normal, alkaline phosphatase ≤ 6 x upper limit of normal For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN; for patients receiving therapeutic anticoagulation: stable anticoagulant regimen.

* Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures.

Exclusion Criteria:

* Patient without neoadjuvant therapy or those who received a neoadjuvant therapy other than FLOT.
* Known hypersensitivity against 5-FU, leucovorin, oxaliplatin, or docetaxel.
* Other known contraindications against, 5-FU, leucovorin, oxaliplatin, or docetaxel.
* Clinically significant active coronary heart disease, cardiomyopathy or congestive heart failure, NYHA III-IV.
* Clinically significant valvular defect.
* Criteria of primary unresectability, e.g.:

Radiologically documented evidence of major blood vessel invasion or invasion of adjacent organs (T4b).

Patients with involved retroperitoneal (e.g. para-aortal, paracaval or interaortocaval lymph nodes) or mesenterial lymph nodes (distant metastases!).

* Other severe internal disease or acute infection.
* Peripheral polyneuropathy ≥ NCI Grade II.
* Patient has undergone major surgery within 28 days prior to enrollment except staging laparoscopy.
* Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or ascites.
* On-treatment participation in another interventional clinical study in the period 30 days prior to inclusion and during the study.
* Patient pregnant or breast feeding, or planning to become pregnant.
* Any other concurrent antineoplastic treatment including irradiation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-10-10 (Estimated); Study Completion 2029-01-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of Overall survival (OS) in both arms | from randomization up to 5 years
  Overall survival (OS) where OS is defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
Comparison of Overall survival rates at 3 and 5 years in both arms | 3 and 5 years after randomization
  Overall survival rates at 3 & 5 years defined as the percentage patients known to be alive after 3 and 5 years referring to the total number of patients randomized into the respective treatment arm
Comparison of progression-/disease-free survival (PFS/DFS) between arms | from randomization up to 5 years
  PFS/DFS is defined as the time from randomization to disease progression or relapse after surgery or death from any cause.
Comparison of peritoneal relapse rate in both arms | from randomization up to 5 years
  Peritoneal relapse rate defined as the percentage of patients with peritoneal relapse referring to the total number of patients randomized into the respective treatment arm
PFS/DFS rates at 2, 3 & 5 years | 2, 3 & 5 years after randomization
  PFS/DFS rates at 2, 3 & 5 years defined as the percentage of patients without disease progression or relapse after surgery or death from any cause after 2, 3 and 5 years referring to the total number of patients randomized into the respective treatment arm
Rate of surgical serious adverse events (SAEs) | After randomization of the patient until 30 days after last study-specific treatment
  Rate of surgical serious adverse events, according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE Version 5.0) grade ≥ 3 adverse events and grade ≥ 3 laboratory toxicities.
Patient reported outcomes: Quality of life EORTC QLQ C30 questionnaire | From date of screening until the date of first documented progression or last visit before date of death from any cause, whichever came first, assessed 8 weeks +/- 7 days until EOT, afterwards every 3 months up to 2 years after last patient in
  The QoL analyses will include QoL mean values, QoL response and time to symptom deterioration (TTSD) defined as the time interval between randomization and the first decrease by ≥ 10-points. All randomly assigned patients with a baseline and at least one post-baseline assessment will be included in TTSD analyses. Patients without observed deterioration will be censored at the time of their last QoL assessment. Questionnaires given to the patients (validated quality of life questionnaires EORTC QLQ C30).
  EORTC QLQ C30 contains 30 questions:
  28 questions regarding body fitness, daily routines, restrictions at work and hobby, appetite, fatigue, cough, breathlessness, pain, tiredness, and body conditions from (1) to (4); 1 (not a bit), 2 (little), 3 (moderate), 4 (much).
  2 questions regarding state of health and Quality of life with a horizontal rating from 1 to 7; 1 (very bad), 7 (excellent).
Patient reported outcomes: VAS pain assessment form | From date of screening until the date of first documented progression or last visit before date of death from any cause, whichever came first, assessed 8 weeks +/- 7 days until EOT, afterwards every 3 months up to 2 years after last patient in
  The patient´s assessment of their current level of pain on a 100-mm horizontal VAS. The left-hand extreme of the line should be described as "no pain" and the right-hand as "unbearable pain".
Rate of post-operative morbidity/mortality at day 30 after surgery acc. to Clavien-Dindo classification | at day 30 after surgery
  Rate of post-operative morbidity/mortality will be assessed at day 30 after surgery acc. to Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zakharenko, PhD, Principal Investigator — First Pavlov State Medical University of St. Petersburg; Ilya Vervekin, Study Chair — First Pavlov State Medical University of St. Petersburg
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.